CLINICAL TRIAL: NCT06360250
Title: Multicenter, Randomized, Blinded, Controlled Phase I / Clinical Trial Evaluating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of the Fully Human Anti-tetanus Toxin Monoclonal Antibody A82 / B86 Injection Combination
Brief Title: Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of the Fully Human Anti-tetanus Toxin Monoclonal Antibody A82 / B86 Injection Combination Formulation
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Changchun BCHT Biotechnology Co. (Industry)
Collaborators: The First Affiliated Hospital of Yunnan University of Traditional Chinese Medicine (Unknown); Anning City First People's Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: B2001-F20220601
Record Dates: First submitted 2024-04-07; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Clostridium Tetanus
Keywords: Monoclonal antibody to tetanus; Safety; tolerability; pharmacokinetics; pharmacodynamics; immunogenicity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group (Experimental): Each dose (1.0 ml) contained 1.25 mg of fully human anti-tetanus toxin monoclonal antibody A82 and 1.25 mg of fully human anti-tetanus toxin monoclonal antibody B86,2.5 mg (1.0 ml) / vial
  Interventions: Drug: Human anti-tetanus toxin monoclonal antibody A82 / B86 injection combination preparation; Biological: Adsorbed tetanus vaccine (TT)
- Positive control group (Active Comparator): Tetanus with human immunoglobulin
  Interventions: Drug: Tetanus human immunoglobulin (HTIG); Biological: Adsorbed tetanus vaccine (TT)
- Placebo group (Placebo Comparator): There were no active ingredients, and other ingredients were the same
  Interventions: Drug: Whole-human anti-tetanus toxin monoclonal antibody A82 / B86 injection placebo; Biological: Adsorbed tetanus vaccine (TT)

INTERVENTIONS:
Drug: Human anti-tetanus toxin monoclonal antibody A82 / B86 injection combination preparation — Each dose (1.0 ml) contained 1.25 mg of human anti-tetanus toxin monoclonal antibody A82 and 1.25 mg of human anti-tetanus toxin monoclonal antibody B86.
  Arms: Experimental group
Drug: Tetanus human immunoglobulin (HTIG) — Tetanus human immunoglobulin (HTIG)
  Arms: Positive control group
Drug: Whole-human anti-tetanus toxin monoclonal antibody A82 / B86 injection placebo — There were no active ingredients, and other ingredients were the same
  Arms: Placebo group
Biological: Adsorbed tetanus vaccine (TT) — containing tetanus toxoid titer not less than 40 IU

SUMMARY:
To evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and immunogenicity of the full human anti-tetanus toxin monoclonal antibody A82 / B86 injection combination formulation

DETAILED DESCRIPTION:
Ia (separate administration phase) To evaluate the safety and tolerability of a single intramuscular injection of different doses of CBL8851 injection in healthy adult Chinese volunteers.

1. To evaluate the pharmacokinetic characteristics of a single intramuscular injection of different doses of CBL8851 injection in Chinese healthy adult volunteers;
2. To evaluate the pharmacodynamic characteristics of a single intramuscular injection of different doses of CBL8851 injection in Chinese healthy adult volunteers;
3. To evaluate the immunogenicity characteristics of a single intramuscular injection of different doses of CBL8851 injection in Chinese healthy adult volunteers.

Ib (Drug interaction phase) To evaluate the safety and tolerability of intramuscular CBL8851 injection combined with tetanus vaccine in Chinese healthy adult volunteers.

1. To evaluate the pharmacodynamic characteristics of the intramuscular CBL8851 injection combined with the adsorption of tetanus vaccine in Chinese healthy adult volunteers, and to evaluate the drug interaction;
2. To evaluate the pharmacokinetic characteristics of intramuscular CBL8851 injection plus tetanus vaccine in Chinese healthy adult volunteers;
3. To evaluate the immunogenicity characteristics of intramuscular CBL8851 injection combined with tetanus vaccine in Chinese healthy adult volunteers.

II designated time Compare the neutralizing antibody activity of intramuscular CBL8851 injection and tetanus human immunoglobulin in Chinese adult volunteers to select the best dose for subsequent efficacy confirmatory tests.

1. to compare the safety of intramuscular CBL8851 injection with tetanus human immunoglobulin in Chinese adult volunteers;
2. To evaluate the immunogenicity characteristics of intramuscular CBL8851 injection in Chinese adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Before the trial, I have a detailed understanding of the nature, significance and possible benefits of the trial, possible inconvenience and potential risks and discomfort, and volunteered to participate in this clinical trial, be able to communicate well with researchers, comply with the requirements of the whole study, and signed a written informed consent;
2. Men or women aged 18~59 (including boundary values) at the time of screening;
3. The weight of female volunteers was 45.0 kg, male volunteers were 50.0 kg, and the body mass index (BMI) was between 18.0 and 27.0 kg / m2 (including the boundary value) (BMI= weight kg / height m2);
4. female volunteers from the 14 days before the first dose to 3 months after the end of the test and voluntary use at least one acceptable contraceptive method, male volunteers from the first time to the trial within 3 months no fertility or donate sperm plan and voluntary use of at least one acceptable contraceptive method.

Exclusion Criteria:

1. People who are known to be allergic to experimental drugs (including excipients and similar drugs), or who suffer from severe allergic diseases or allergies (such as allergic to two or more drugs, food or pollen), may damage the safety of the volunteers by the judgment of the investigator (inquiry);
2. Those with a clear history of allergy to essential substances (such as skin disinfectants and alcohol substances that may be exposed to) during the test (inquiry);
3. tetanus vaccine or tetanus toxin antigen component (DPT vaccine, DPT vaccine, meningitis conjugate vaccine, etc.) vaccinated in the previous 10 years (inquiry);
4. Those who received any live attenuated vaccine or inactivated vaccine (including COVID-19 vaccine) within 1 month (30 days) before the first dose, or received the above vaccine within 3 months after the planned dose (inquiry);
5. Previous history of tetanus infection (inquiry);
6. Known or suspected immune deficiency (inquiry), including immunosuppressive therapy (radiation therapy, chemotherapy, corticosteroid hormones, antimetabolism, cytotoxic drugs) (inquiry, inquiry), HIV infection (inquiry) within 3 months before the first dose (90 days);
7. History of active infection or disease with one of the following conditions:

   Systemic systemic anti-infective therapy within 14 days before the first administration (inquiry, inquiry); Recurrent, chronic, or other active infections, as assessed by the investigator, may increase the volunteer risk (inquiry).
8. Patients with chronic diseases (including hypertension, diabetes, hyperlipidemia, hyperuricemia, etc.) (phase I only); chronic diseases (including hypertension, diabetes, hyperlipidemia, hyperuricemia, etc.) and unstable control (phase II only) (inquiry);
9. People with a history of tuberculosis who are not cured or have active tuberculosis infection during screening (inquiry);
10. has a history of malignancy (active or has been treated but not clearly clinically cured, or may recur during the trial) (inquiry);
11. Patients with a previous history of convulsions, epilepsy, mental or neurological system, or a family history of convulsions or epilepsy (inquiry);
12. Those who have a history of clinically serious disease within 6 months before the first dose (180 days) and are not cured, or those who have acute or chronic diseases that may significantly affect the in vivo process or safety evaluation of the investigational drug (inquiry, inquiry);
13. Those who had received major surgery within 3 months (90 days) prior to the first dose, or who may have significantly affected the process or safety evaluation of the study drug, or who planned to undergo surgery during the study (inquiry, inquiry);
14. Those who have been used or are in significant impact on the in vivo process or safety evaluation of the investigational drug (inquiry, inquiry);
15. Use of other clinical trial drugs / devices within 3 months (90 days) prior to the first dose, or <5 clearance half-lives since the last dose of previous experimental drugs (whichever is older), or participation in other clinical trial planners during the trial (inquiry, inquiry);
16. Drinking more than 28 units of alcohol per week (1 unit =285 ml beer or 25 ml spirits or 40% alcohol) for 3 months (90 days) before the first dose (inquiry);
17. Smoking more than 10 cigarettes or equal amounts of tobacco per day for 1 month (30 days) prior to the first dose (inquiry);
18. Blood loss / blood donation over 400 ml (except female physiologic blood loss) within 3 months (90 days) before the first dose, or receiving blood transfusion or using blood products, or planned to donate during the trial or within 1 month (30 days) after the end of the trial (inquiry);
19. Patients with positive rapid IgG during the screening period (examination);
20. Those with a history of substance abuse (inquiry) or those positive for substance abuse screening during the screening period (examination);
21. Hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), hepatitis C antibody (HCV-Ab) antibody, Treponema syphilis antibody (TPPA) or antibody to human immunodeficiency virus (Anti-HIV);
22. Ear temperature during the screening period is> 37.5℃ (examination);
23. Physical examination, vital signs (blood pressure, pulse rate), electrocardiogram, other laboratory tests (laboratory tests not listed separately) or other auxiliary test results during the screening period are judged as abnormal and clinically significant by the study doctor (examination);
24. Women in pregnancy or lactation (inquiry) or those with a positive pregnancy test (examination);
25. Patients with a history of needle acupuncture, blood halo (inquiry), unable to tolerate or without adequate venous access to allow regular venipuncture (inquiry, examination);
26. The volunteers may be unable to cooperate with the study for other reasons or the investigators is not unsuitable for inclusion.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 190 (Estimated)
Dates: Start 2024-04-10 (Estimated); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Safety evaluation index | Twelve months
  All observed adverse events, serious adverse events, including but not limited to: Clinical indicators Physical examination; vital signs; 12-lead ECG; local reaction; systemic reaction. Laboratory tests: blood routine, urine routine, blood biochemistry (liver function, kidney function, fasting blood glucose, blood lipid, myocardial enzyme spectrum, electrolytes), blood coagulation routine, blood / urine pregnancy test (only fertility women), etc.; Other auxiliary examinations: chest CT and abdominal B-ultrasound.

SECONDARY OUTCOMES:
PK evaluation index | Twelve months
  Peak Plasma Concentration (Cmax)
PK evaluation index | Twelve months
  Area under the plasma concentration versus time curve (AUC)
PK evaluation index | Twelve months
  Maximum peak time (Tmax)
PK evaluation index | Twelve months
  Half-life period(T1/2)
PK evaluation index | Twelve months
  MeanResidenceTime（MRT）
PK evaluation index | Twelve months
  Apparent clearance rate (CL / F)
PD evaluation index | Twelve months
  The level of neutralizing antibodies against tetanus toxin at 6 h, 12 h, and 24 h, on days 2,3,7,14,21,28,42,56,84, and 105
PD evaluation index | Twelve months
  6 h, 12 h, and 24 h at days 2,1,2,3,7,14,21,28,42,56,84, and 105 (0.01 IU / ml [modified ligand binding assay] or 0.1 IU / ml [direct ligand binding assay])
PD evaluation index | Twelve months
  Duration of 0.01 IU / ml (modified ligand binding assay) or 0.1 IU / ml (direct ligand binding assay) at days 2,3,7,24,21,56,84 and 24 h after administration
Immunogenicity evaluation index | Twelve months
  Positive rate of anti-drug antibody (ADA) and neutralizing antibody (Nab) on days 7,14,28,56, and 105 of CBL8851 injection (CBL8851A82 and CBL8851B86).